CLINICAL TRIAL: NCT07206771
Title: Knowledge, Attitudes, and Practices Among Parents of Children With Napkin Dermatosis and Its Patterns in Assiut University Hospitals
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Donia Ahmed zakaria, doctor, Assiut University
Other Study IDs: napkin dermatosis
Record Dates: First submitted 2025-09-26; First posted 2025-10-03 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Napkin Dermatosis
Keywords: knowledge of napkin dermatosis; pattern of napkin skin lesion

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluate the level of knowledge , attitude and practices among parents of children with napkin dermatosis and assess the pattern of napkin dermatosis among children up to 2 years old attending Assiut University Hospital (AUH).

DETAILED DESCRIPTION:
Napkin dermatosis, commonly referred to as diaper rash or napkin dermatitis, is a frequent inflammatory skin condition affecting the diaper area of infants and young children, particularly under three years of age [1,2]. It is characterized by erythematous macules, papules, and sometimes erosions or secondary infections. Prevalence rates vary between 4% and 35%, with peak incidence between 8 and 12 months [1-3].Multiple factors contribute to its development, including prolonged exposure to moisture, urine, and feces, which compromise the skin barrier and increase susceptibility to irritants and infections. Interaction of urine with skin bacteria produces ammonia, raising skin pH and promoting irritation [4,5]. Introduction of solid foods can further exacerbate inflammation, and secondary infections, particularly by Candida albicans, may complicate the clinical course [6,7].Caregivers' knowledge, attitudes, and practices are critical in preventing and managing napkin dermatosis. Frequent diaper changes, use of barrier creams, and avoiding irritant products significantly reduce its risk [8-9].Parental knowledge and awareness about proper diaper care, prevention strategies, and early recognition of complications play a pivotal role in reducing the incidence and severity of napkin dermatosis [7]. However, evidence suggests that parental awareness and adherence to recommended practices vary widely, especially in regions lacking structured educational programs [10,11].the rationale for this study is to assess Parental knowledge, attitudes, and practices, and describe the patterns of napkin dermatosis among children attending Assiut University Hospitals, ultimately improving child health and parental care behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Children aged up to 2 years attending Assuit University Chlidren's Hospital and dermatology outpatient clinics in AUH during the study period , presenting with skin changes in the diaper area.
* Children whose parents and caregivers provide informed consent for participation.

Exclusion Criteria:

* parents and caregivers who refuse or are unable to give informed consent.
* Infants on admission , severely ill or immunocompromised

Ages: 1 Day to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 0-24 months presenting with napkin dermatosis at Assiut University Hospitals outpatient dermatology and pediatric clinics
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
parental knowledge ,attitude and practice regarding napkin dermatosis | At baseline (during recruitment,within study period)
  the level of knowledge ,attitude and practice of parents and caregivers regarding causes, prevention, and management of napkin dermatosis, expressed as a composite knowledge score obtained from the questionnaire
Rate and pattern of napkin dermatosis among children up to 2 years attending Assiut University Hospital | Within 12 months of study enrollment
  Distribution and frequency of clinical types of napkin dermatosis (e.g., irritant contact dermatitis, candidiasis, bacterial infections, seborrheic dermatitis, etc.).

SECONDARY OUTCOMES:
Correlation between parental awareness and severity of napkin dermatosis | At the end of the study (12 months)
  Statistical association between caregivers' knowledge, attitude, and practice (KAP) scores and the clinical severity/type of napkin dermatosis in their children.
Identification of socio-demographic and clinical risk factors | Within 12 months of study enrollment.
  Analysis of potential risk factors for napkin dermatosis, including socio-demographic variables (parental education, income, etc.) and clinical factors (diarrhea, diaper type, hygiene practices)
Frequency of secondary infections associated with napkin dermatosis | Within 12 months of study enrollment
  Measurement of occurrence of secondary bacterial or fungal infections complicating napkin dermatosis in affected children.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://doi.org/10.31579/2578-8949/149
- See also: Related Info — https://doi.org/10.4094/chnr.2019.25.2.112